CLINICAL TRIAL: NCT05296343
Title: Developing Guidelines for Parental Involvement in the Emergency Care of Suicidal Adolescents and Young Adults: a Qualitative Study
Brief Title: Guidelines for Parental Involvement in the Care of Suicidal Youth
Acronym: S-Urg-Quali
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: AOI 2021 LACHAL; 2021-A03244-37 (Other: ANSM)
Record Dates: First submitted 2022-03-14; First posted 2022-03-25 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Suicide, Attempted; Emergencies
Keywords: Adolescent; Parent; Qualitative study; Guidelines
MeSH Terms: conditions — Suicide, Attempted; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents and young adults: Boys and girls from 15 to 25 years old admitted to an Emergency Department (ED) following a suicidal act or considered as such by the medical team
- Parents: One or the two parents of the included adolescents and young adults
- Healthcare professionals: Professionals working in one emergency departments of the inclusion centers and who usually take care of suicidal adolescents and young adults

SUMMARY:
Parents occupy a central place in the emergency care of suicidal adolescents and young adults. However, from 15 to 25yo, three different administrative situations exist in France:

* <16yo: admission to a child ED by a team trained to receive the youngest patients.
* 16-18yo: admission to an adult ED by team devoted to adult care, no exit without parents' authorization.
* >18yo: admission to an adult ED by team.

Laying on qualitative observational protocol and a Delphi approach, this study will explore the perspective of adolescents and young adults following a suicidal attempt, the perspective of their parents, and the perspective of their healthcare professionals to build guidelines for parental involvement in care of suicidal youths.

DETAILED DESCRIPTION:
Suicide is the second leading cause of death among 15-25 year olds, with the highest rate of hospitalization for SC of any age group. The psychopathology of suicidal behavior in adolescents and young adults (AYA) is homogeneous: risk factors, precipitating factors, representations. Parents occupy a central place in care. They are i) involved in the care decision; ii) actively involved in care; and ii) a source of motivation for trust and adherence to care.

However, if the psychopathology of suicidal crisis is homogeneous, the transition between pediatric and adult care implies very different management in the emergency department (ED). In France, three situations can be described:

* <16yo: admission to a child ED by a team trained to receive the youngest patients.
* 16-18yo: admission to an adult ED by team devoted to adult care, no exit without parents' authorization.
* >18yo: admission to an adult ED by team devoted to adult care, no right to contact the parents in case of patient opposition.
* Before 16 years of age: admission to the children's UAS, care by a team trained to receive the youngest patients.
* 16-18 years: admission to the adult UAS, care by adult professionals, clinical and legal particularities of care for minors.
* After 18 years old: admission to adult UAS, legal constraints of the adult care setting.

The objectives of this qualitative observational study is to build guidelines for the involvement of the parents in the care in these three situations.

The study will include adolescents and young adults from the three situations, their parents and the professionals who take care of them. Individual semi-structured interviews will be organized to collect their experiences. Qualitative analyses will be conduct, following Interpretative Phenomenological Analysis. A pre-approved guideline will be construct and a Delphi approach will be conducted to approved the final version of the guideline.

ELIGIBILITY:
Inclusion Criteria:

Adolescents and Young adults

* Admitted to an Emergency Department (ED) following a suicidal act or considered as such by the medical team

Parents

* Parents of the included youths >18y

Healthcare professionals

* >18y
* Working in ED
* Usually taking care of suicidal youths

All the participants

* French speaking
* Affiliation to a social security regime
* Participation agreement

Exclusion Criteria:

All the participants

* Present an acute somatic or psychiatric disease which may hinder the well organization of the interview

Ages: 15 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Any adolescent and young adult admitted to an Emergency Department (ED) in one of the inclusion center following a suicidal act or considered as such by the medical team. Their parents; healthcare professionals working in ED of the inclusion centers.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Developing guidelines defining the role of parents in the medical decision and the care of the youths | Day 1
  Thematic framework summarizing the perspectives of three groups of participants.

SECONDARY OUTCOMES:
Describing each context of care | Day 1
  Qualitative description of each of the three context of care (<16y, 16-18y, >18y)
Describing expectations from each group | Day 1
  Qualitative description of each of the three participant groups (adolescents and young adults, parents, professionals)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lachal, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France